CLINICAL TRIAL: NCT00297934
Title: Influence of Instrument-Applied Spinal Manipulative Therapy on Dual-Task Performance Involving Complex Postural and Cognitive Tasks
Brief Title: Spinal Manipulative Therapy: Dual-Task Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCC-06-02
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2006-10

CONDITIONS: Balance
Keywords: dual-task; postural control; cognitive

INTERVENTIONS:
Device: Pro-adjuster mechanical spinal manipulative device

SUMMARY:
The purposes of this study is to determined the effects of instrument applied spinal manipulative therapy upon dual-task performance involving complex postural and cognitive task.

DETAILED DESCRIPTION:
This study sought to determine whether a 2-week regimen of spinal manipulative therapy could improve postural control under 2 conditions. Condition one was a complex postural task which consisted of a shoulder width stance on a compliant surface with eyes closed to remove visual input. Condition 2 was as above with the addition of visio-spatial cognitive task (serial 7s subtraction). These tasks were performed on a force-place designed to capture center of pressure data. Data was captured prior to the onset of therapy and then again after 6 treatment sessions (2-week period). Data was also collected 1 week post treatment to note any lasting effects following therapy. This pilot study utilized a repeated measures designed with no control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants

Exclusion Criteria:

* No injuries
* No surgeries
* No visual, vestibular, or somatosensory disorders capable of affecting balance

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2006-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Sway velocity using a NeuroCom Balance Master Forceplate

CONTACTS AND LOCATIONS:
Overall Officials: Rodger Tepe, PhD, Study Director — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States